CLINICAL TRIAL: NCT04499755
Title: Efficacy of Nucleo CMP Forte in Traumatic Brain Injury in Pediatrics: A Randomized Controlled Trial
Brief Title: Efficacy of Nucleo CMP Forte in Traumatic Brain Injury in Pediatrics
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KFS protocol
Record Dates: First submitted 2020-08-01; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nucleo CMP forte (Experimental): Nucleo CMP forte twice daily for 6 weeks with supportive treatment.
  Interventions: Drug: Nucleo CMP Forte
- Supportive treatment (No Intervention): Supportive treatment only.

INTERVENTIONS:
Drug: Nucleo CMP Forte — Nucleo CMP Forte twice daily for 6 weeks
  Other Names: Nucleoforte
  Arms: Nucleo CMP forte

SUMMARY:
Efficacy of Nucleo CMP Forte in Traumatic Brain Injury in Pediatrics

DETAILED DESCRIPTION:
The study aims to study the Efficacy of Nucleo CMP Forte in Traumatic Brain Injury in Pediatrics

ELIGIBILITY:
Inclusion Criteria:

* Children with traumatic brain injury: Moderate and Severe.

Exclusion Criteria:

* Underlying CNS disorders,

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with improved glasgow coma score | 2 months
  The number of patients with improved glasgow coma score

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Salamah, Lecturer, Principal Investigator — Pediatrics department - Kafr-Elsheikh University; Mohamed Elbahnasawy, lecturer, Principal Investigator — Emergency Department- Tanta University.
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No